CLINICAL TRIAL: NCT05090852
Title: High Velocity Nasal Insufflation (Hi-VNI) Use in Upper Airway Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natasha Mirza (Other)
Responsible Party: Sponsor-Investigator, Natasha Mirza, Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 834412
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Upper Airway Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hi-VNI as primary or adjunct oxygenation technique (Experimental): Hi-VNI used as a primary or adjunct oxygenation technique during upper airway surgery
  Interventions: Device: Hi-VNI

INTERVENTIONS:
Device: Hi-VNI — Hi-VNI used instead of or along with endotracheal intubation or jet ventilation to provide oxygen to patients during upper airway surgery

SUMMARY:
The goals of this study are to establish the efficacy of Hi-VNI (High Velocity Nasal Insufflation) in upper airway surgery from the anesthesiologist's and surgeon's perspectives, and to describe the ideal patient and the ideal pathology as well as suitable clinical scenarios when this oxygenation technique should be selected.

DETAILED DESCRIPTION:
The most challenging aspects of laryngeal and laryngotracheal procedures are difficulty of exposure and airway management. These procedures require use of microlaryngeal instruments through a small lumen of a rigid laryngoscope, and are oftentimes difficult to perform with a standard endotracheal tube in place. Similarly, when performing endoscopic evaluation of the trachea, access to the space and visualization of the entire 360-degree view of the trachea is crucial.

To overcome these challenges, a number of techniques for oxygen delivery have evolved over time. Among them are use of a small endotracheal tube, use of jet ventilation and intermittent apnea with periodic removal of the endotracheal tube. The aforementioned methods of airway management carry inherent risks of airway injury, can be accompanied by brief periods of hypoxia or hypercarbia, and can sometimes lead to tenuous airway management scenarios for both the surgeon and the anesthesiologist when clear communication and familiarity with the airway management plan during the procedure are sub-optimal. For this reason, there is an ongoing search for acceptable solutions to minimize these risks during upper airway surgery.

One of the newly emerging advanced oxygenation techniques, also known as Hi-VNI (High Velocity Nasal Insufflation), allows for delivery of humidified oxygen through a specialized high-flow nasal cannula at rates of up to 40 l/min. This non-invasive high flow respiratory support system is currently being used in the treatment of respiratory failure in both adult and pediatric patients. This technique provides sustained oxygenation due to reduction in airway resistance, a build-up of airway pressure with oxygen-rich gas and active gas exchange, which lead to flushing of anatomic dead space, and delivery of oxygen into the lungs. This oxygenation technique can be used both in spontaneously breathing patients and under apneic conditions, while providing an unobstructed surgical view with the glottis, subglottis and trachea fully accessible for instrumentation.

The goal of this study is to establish the efficacy of Hi-VNI in upper airway surgery, to document the advantages and disadvantages of this technique from the standpoint of the airway surgeon and the anesthesiologist, and to provide more information about the optimal patient and airway pathology as well as suitable clinical scenarios when Hi-VNI device can be used for oxygenation during upper airway surgery. The researchers hypothesize that in appropriate clinical situations, Hi-VNI can ease airway management, shorten case duration, and provide superior operating conditions including space for instrumentation during upper aerodigestive tract procedures.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective upper airway surgery at the University of Pennsylvania

Exclusion Criteria:

* Underlying medical conditions in which brief periods of hypoxemia or hypercarbia are not well tolerated
* Coronary artery disease
* Severe heart failure with EF < 40% or implanted ICD
* Pulmonary hypertension or pulmonary fibrosis
* History of increased intracranial pressure
* History of skull base or intracranial surgery
* Severe nasal obstruction
* Extremely low or extremely high BMI (BMI <16 or >40)
* At high risk for aspiration
* Taken to OR for urgent or emergent upper airway surgery

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Mirza, MD, Principal Investigator — Department of Otorhinolaryngology - Head and Neck Surgery
Locations (1):
- Hospital of the University of Pennsylania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hi-VNI as Primary or Adjunct Oxygenation Technique
Started | 31
Completed | 26
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: Patients undergoing anesthesia for airway laryngeal surgery
Groups:
- Hi-VNI as Primary or Adjunct Oxygenation Technique: Hi-VNI used as a primary or adjunct oxygenation technique during upper airway surgery
  Hi-VNI used instead of or along with endotracheal intubation or jet ventilation to provide oxygen to patients during upper airway surgery
Arm/Group | Hi-VNI as Primary or Adjunct Oxygenation Technique
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 1
  Unknown or Not Reported | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Surgical Case Completion Rate Using HVNI With or Without Converting to Alternative Mode of Oxygenation
Description: For each case, the ability to complete the surgical procedure with use of only Hi-VNI device for oxygenation will be assessed.
  Patients were oxygenated with Hi-VNI at a flow rate of 40 L/min and FiO2 of 100%. Patients with spO2 < 93 or TcCO2 > 65 during the procedure were converted to an alternative means of oxygenation, including mask ventilation and endotracheal intubation.
  The primary outcome measure is the surgical case completion rate with or without converting to alternate means of oxygenation.
Time Frame: 1 day
Population: Adult patients undergoing upper airway surgery who received HVNI, We compared patients who successfully completed their anesthesia for the surgical case with HVNI vs patients who had to be intubated.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With HVNI and Patients With Intubation: Patients who completed their anesthesia with HVNI and patients who were switched to intubation
Arm/Group | Patients With HVNI and Patients With Intubation
Number analyzed (Participants) | 31
Participants
  Total number of patients who successfully received HVNI only | 19
  Number of patients who received HVNI and also required conversion to alternate oxygenation | 7
  Number of patients who were enrolled but did not receive HVNI | 5

ADVERSE EVENTS:
Time Frame: 24 hours after the start of case
Groups:
- Patients With HVNI and Patients With Intubation: There were no adverse events reported for patients in either group.
Arm/Group | Patients With HVNI and Patients With Intubation
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT05090852/Prot_SAP_000.pdf